CLINICAL TRIAL: NCT04541485
Title: Phase I Study to Evaluate the Safety, Tolerability, and Pharmacodynamics (PD) of DWRX2003 (Niclosamide IM Depot) Injection Following Intramuscular Administration in COVID-19 Patients
Brief Title: To Evaluate Safety, Tolerability and Pharmacodynamics of DWRX2003 Against COVID-19 (in Philippines)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrolment was suspended since 09Dec2020 due to a lack of COVID-19 patients.
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1516101_Phillipphines
Record Dates: First submitted 2020-09-07; First posted 2020-09-09 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: COVID-19 Patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental: Cohort 1 (96 mg) (Experimental): 24 mg/0.1 mL x 4 sites
  Interventions: Drug: DWRX2003; Drug: Placebo
- Experimental: Cohort 2 (288 mg) (Experimental): 72 mg/0.3 mL x 4 sites
  Interventions: Drug: DWRX2003; Drug: Placebo
- Experimental: Cohort 3 (480 mg) (Experimental): 120 mg/0.5 mL x 4 sites
  Interventions: Drug: DWRX2003; Drug: Placebo
- Experimental: Cohort 4 (672 mg) (Experimental): 168 mg/0.7 mL x 4 sites
  Interventions: Drug: DWRX2003; Drug: Placebo
- Experimental: Cohort 5 (960 mg) (Experimental): 240 mg/1.0 mL x 4 sites
  Interventions: Drug: DWRX2003; Drug: Placebo

INTERVENTIONS:
Drug: DWRX2003 — Intramuscularly injection at pre-defined injection sites
Drug: Placebo — Intramuscularly injection at pre-defined injection sites

SUMMARY:
This study is designed to assess the safety and tolerability of single doses of DWRX2003 in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 65 years of age, inclusive at time of signing the ICF.
2. Subjects with low to moderate risk defined as NEWS COVID-19 infection as confirmed by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) assay 72 hours prior to clinical trial enrollment.

Exclusion Criteria:

1. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee). Please note patients with allergies which can be managed without treatment can be included based on the decision of the Investigator (or designee).
2. Significant history, clinical manifestation of any medical disorder or any comorbid conditions which in the opinion of the investigator may interfere with the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | follow-up 42 days after dosing
  Incidence, severity and causality of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Time to SARS-CoV-2 eradication (days) by Nasopharyngeal specimen | follow-up 42 days after dosing
Rate of SARS-CoV-2 eradication by Nasopharyngeal specimen | at Day 3, 7, 10 and 14

CONTACTS AND LOCATIONS:
Locations (1):
- Deawoong pharmaceutical, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No